CLINICAL TRIAL: NCT04444765
Title: Hemodynamic and Respiratory Tolerance of Intermittent Hemodialysis (Acetate Free Biofiltration and Bicarbonate-based Intermittent Dialysis) in Critically Ill Patients
Brief Title: Hemodynamic and Respiratory Tolerance of Intermittent Hemodialysis in Critically Ill Patients
Acronym: COOBrA
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/19/0496
Record Dates: First submitted 2020-05-29; First posted 2020-06-24 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; renal replacement therapy; acetate free biofiltration; bicarbonate-based hemodialysis; C02 removal; intensive care unit; critical care
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with bicarbonate-based intermittent dialysis: Dialysate is composed by electrolytes, including calcium, and bicarbonate. To avoid calcium carbonate precipitation, dialysate has to be supplemented with acids (citric acid, chloride acid or acetic acid).
  Interventions: Other: Collection of clinical and biological data during renal replacement therapy sessions
- Patients with acetate free biofiltration dialysis: Acetate free biofiltration (AFB-K)is a technique that does not require dialysate acidification
  Interventions: Other: Collection of clinical and biological data during renal replacement therapy sessions

INTERVENTIONS:
Other: Collection of clinical and biological data during renal replacement therapy sessions — Collection of clinical and biological data during renal replacement therapy sessions. Two additional blood samples collected during and after RRT session (critically ill patients all have arterial catheter thus additional samples will not need additional puncture).

SUMMARY:
Acute kidney injury (AKI) affects up to 30% of critically ill patients and is associated with increased rates of mortality. Up to 60% of patients with AKI will ultimately require renal replacement therapy (RRT). Intermittent hemodialysis (IHD) is one of the main methods of RRT worldwide. In IHD-bicar, dialysate is composed by electrolytes, including calcium, and bicarbonate. To avoid calcium carbonate precipitation, dialysate has to be supplemented with acids (citric acid, chloride acid or acetic acid). However, IHD-bicar may be associated with hemodynamic instability or respiratory intolerance, mainly related to the CO2 release in the circulation during IHD (HCO3- <--> CO2 + H2O). Some recent studies showed that acetate free biofiltration (AFB-K), a technique that does not require dialysate acidification, could be associated with better hemodynamic stability and to a lower amount of CO2 delivered to the patients. AFB-K may thus improve the hemodynamic and respiratory tolerance of intermittent RRT in critically ill patients.

DETAILED DESCRIPTION:
In this prospective observational study, investigators aim to characterize the hemodynamic and respiratory tolerances of HDI-bicar and AFB-K in critically ill patients requiring RRT.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Invasive monitoring of blood pressure
* Non opposition to the research
* Admission to the intensive care unit
* Need of intermittent hemodialysis

Exclusion Criteria:

* Sodium bicarbonate infusion
* Pregnancy or breastfeeding
* Juridical protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute kidney injury
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Occurence of hemodynamic event | From admission to discharge, up to 4 hours
  The occurrence of at least one of the following events will be considered a hemodynamic event :
  * Hypotension (decrease of systolic or mean blood pressures ≥ 15 and ≥ 10% respectively)
  * Tachycardia (increase of heart beating ≥ 20%)
  * Cardiac arrythmia (junctional tachycardia, atrial fibrillation, flutter, ventricular tachycardia or fibrillation)
  * Decrease of the cardiac output ≥ 15% (only in patients with invasive cardiac output monitoring)
  * Starting (or increase dosing) of norepinephrine ≥ 0.1 µg/kg/min

SECONDARY OUTCOMES:
Change in maximal PaCO2 | 1 hour after the beginning of dialysis , up to 4 hours
  Evaluation of PaCO2 by arterial blood gas test
Maximum difference of tcPCO2 and etCO2 | From admission to discharge, up to 4 hours
  Evaluation of TcPCO2 and etCO2 by trans-cutaneous measurement
Change in the "strong ion difference" | baseline, 4 hours
  Evaluation of the "strong ion difference" by blood ionogram
Change in plasma pH | 1 hour after the beginning of dialysis session, up to 4 hours
  Evaluation of plasma pH by blood ionogram

CONTACTS AND LOCATIONS:
Overall Officials: Stanislas Faguer, MD, Principal Investigator
Locations (1):
- Hôpital Rangueil, Toulouse, France